CLINICAL TRIAL: NCT04821206
Title: PANLAR's Latin American Registry of Rheumatic Patients Treated With Jak Inhibitors
Acronym: PREJAK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liga Panamericana de Asociaciones de Reumatologia (PANLAR) (Other)
Responsible Party: Principal Investigator, Nicolas Marin Zucaro, MD, Liga Panamericana de Asociaciones de Reumatologia (PANLAR)
Other Study IDs: 5858
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondyloarthritis
Keywords: Rheumatoid Arthritis; Psoriatic Arthritis; Spondyloarthritis; Janus Kinase Inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis | interventions — Antirheumatic Agents; Janus Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Patients with diagnosis of RA, PsA and SpA
  Interventions: Drug: JAK Inhibitor
- Controls: Patients with diagnosis of RA, PsA and SpA
  Interventions: Drug: DMARDs; Drug: biologic DMARDs

INTERVENTIONS:
Drug: DMARDs — New Initiation of a DMARDs
  Groups: Controls
Drug: biologic DMARDs — New Initiation of a biologic DMARDs
  Groups: Controls
Drug: JAK Inhibitor — New Initiation of a JAK Inhibitor
  Groups: Cases

SUMMARY:
This prospective, non-interventional, research registry is designed to study the comparative safety and comparative effectiveness of approved Jak Inhibitors treatment for RA-PsA-SpA in a cohort of patients and theirs controls cared for by rheumatologists across Latin América (LA).

DETAILED DESCRIPTION:
There is scarce data on the real-world safety and effectiveness of Jak in Latin America. This registry will provide reliable data on the use of JAKi in LA, as will be a prospective study involving carefully selected rheumatologists and centers. Soon, a good number of copies of original JAKi will be available in LA, and it is important to keep track of the safety and effectiveness of this drugs in the real world.

The primary objective of the registry is to prospectively study the comparative safety and comparative effectiveness of approved Jak Inhibitors treatment for RA-PsA-SpA in a cohort of patients and theirs controls cared for by rheumatologists across Latin América (LA).

The registry will be a cohort study where cases will be patients with RA, PsA and SpA initiating any approved JAK inhibitor. To have an active control group, patients with RA, PsA o SpA initiating any other disease modifying antirheumatic drug (DMARD) (biologic or not biologic) will also be included in the registry.

It will be a Web based registry, where the investigators will include data related to the cases and controls. Data collected will include, demographics, disease characteristics, disease activity, past and current medications, comorbidities. At each visit adherence with the medications, adverse events, changes in medications, disease activity and disability will be assessed.Patients will be followed up at three months intervals, after inclusion in the registry and thereafter every 6 months during the next three years. Adverse events could be included at any time between visits if the investigator is notified.

ELIGIBILITY:
To be eligible for enrollment into the PREJAK Registry, a patient must satisfy all of the inclusion criteria and none of the exclusion criteria listed below.

Inclusion Criteria

The patient must be:

1. One of the following:

   1. Diagnosis with rheumatoid arthritis (RA) and initiating (prescribed or starting) a Januse Kinase inhibitors (JAKi) for the treatment of RA at the enrollment visit.
   2. Meet the ASAS criteria for axial spondyloarthritis (AxSpA), including radiographic or non-radiographic, and initiating (prescribe or starting) a JAKi for the treatment of AxSpA at the enrollment visit.
   3. Diagnosis with psoriatic arthritis (PsA) and initiating (prescribed or starting) a Januse Kinase inhibitors (JAKi) for the treatment of PsA at the enrollment visit.
2. At least 18 years age or older
3. Able and willing to provide written consent

Exclusion Criteria:

Patients who do not wish to participate or are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will be a cohort study where cases will be patients with RA, PsA and AS initiating any approved JAK inhibitor. To have an active control group, patients with RA or PsA initiating any other disease modifying antirheumatic drug (DMARD) (biologic or not biologic) will also be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of severe adverse events per each one of the drugs included. | 12 months
Incidence rate of severe adverse events per each one of the drugs included. | 24 months
Incidence rate of severe adverse events per each one of the drugs included. | 36 months

SECONDARY OUTCOMES:
Incidence rate of all adverse events for each one of the drugs included. | 12 months
Incidence rate of all adverse events for each one of the drugs included. | 24 months
Incidence rate of all adverse events for each one of the drugs included. | 36 months
Incidence rate of severe infections for each one of the drugs included. years. | 12 months
Incidence rate of severe infections for each one of the drugs included. years. | 24 months
Incidence rate of severe infections for each one of the drugs included. years. | 36 months
Proportion of patients still on each one of the drugs included. | 12 months
Proportion of patients still on each one of the drugs included. | 24 months
Proportion of patients still on each one of the drugs included. | 36 months
Proportion of patients on remission (according to definition) for each one of the drugs included and for each one of the diseases included. | 12 months
Proportion of patients on remission (according to definition) for each one of the drugs included and for each one of the diseases included. | 24 months
Proportion of patients on remission (according to definition) for each one of the drugs included and for each one of the diseases included. | 36 months
Proportion of patients receiving each one of the drugs included and for each one of the diseases included as first, second, third- and fourth-line therapy. | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Hospital Italiano de Buenos Aires, CABA, Buenos Aires
  - Nicolas Marin Zucaro, Ciudad Autonoma Buenos Aires, Buenos Aires

IPD SHARING:
Plan to Share IPD: No